CLINICAL TRIAL: NCT02435563
Title: Dose Adaptation to Offset the Pharmacokinetic Interaction Between Ticagrelor and Ritonavir in Healthy Volunteers by Population-based PK Modeling (Simcyp®)
Brief Title: Dose Adaptation to Offset the Interaction Between Ticagrelor and Ritonavir by Population-based PK Modeling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jules Desmeules, Dr, University Hospital, Geneva
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 13-182
Record Dates: First submitted 2014-09-15; First posted 2015-05-06 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Anti-HIV Agents; cardiovascular agents; drug interactions
MeSH Terms: interventions — Ticagrelor; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor 180 mg (Experimental): Single dose of 180mg ticagrelor administered orally
  Interventions: Drug: ticagrelor 180 mg administrated alone
- Ticagrelor adjusted dose+ritonavir 100mg (Experimental): adpated dose of ticagrelor calculated after PK modelisation with the Simcyp® simulator administered simultaneously with 100 mg ritonavir
  Interventions: Drug: Ticagrelor adjusted dose + ritonavir 100mg

INTERVENTIONS:
Drug: ticagrelor 180 mg administrated alone
  Arms: Ticagrelor 180 mg
Drug: Ticagrelor adjusted dose + ritonavir 100mg
  Arms: Ticagrelor adjusted dose+ritonavir 100mg

SUMMARY:
Ticagrelor is a new generation antiplatelet agent with higher efficacy as compared to clopidogrel and prasugrel in treatment of patients with moderate and high ischemic risks. Ticagrelor is active as such and its hepatic metabolism by CYP3A generates also an active metabolite. Because of the remarkable progress in HIV therapies the number of older age patients is on the rise, requiring adequate cardiovascular treatment. Since frontline HIV therapies include ritonavir, a strong inhibitor of CYP3A enzyme, ticagrelor is contraindicated in these patients because of the expected interaction and bleeding risk. A lower efficacy of clopidogrel and prasugrel, which are both pro-drugs, in the presence of ritonavir has been already demonstrated. Therefore, administration of a lower dose of ticagrelor may be a good alternative in HIV patients in order to lessen the impact of this pharmacokinetic interaction. The aim of this study is to adjust the dose of ticagrelor in case of co-treatment with ritonavir to achieve the same pharmacokinetic profile as administered alone using a physiologically-based pharmacokinetic (PBPK) model.

As the first step, a pharmacokinetic (PK) model for ticagrelor and its active metabolite will be created based on available in vitro and in vivo parameters in healthy volunteers.

An open-label, 2 sessions cross over study will be conducted with 20 healthy male volunteers at Clinical Research Center (CRC) of Geneva University Hospitals (HUG). During the first session of the clinical trial, a single dose 180 mg ticagrelor will be administered to the volunteers and obtained pharmacokinetic data will be fitted into the model for optimization. Thereafter a simulated trial by the Simcyp® simulator in presence of a single dose 100 mg ritonavir will allow evaluating the impact of CYP3A inhibition on the concentration-time profile of ticagrelor and its active metabolite. The necessary dose of ticagrelor to minimize the magnitude of this interaction will be calculated. This new dose will be co-administered with ritonavir in the same volunteers during the second session of the clinical trial. The purpose is to obtain the same PK profile with single dose of 180 mg ticagrelor administered alone and with an adapted dose of ticagrelor co-administered with a single dose 100 mg ritonavir. Moreover, the pharmacodynamic effect of ticagrelor will be measured in both sessions of the clinical trial using two specific platelet function tests: the VAsodilator-Stimulated Phosphoprotein assay (VASP) and VerifyNow® P2Y12. With the same PK profile, the same pharmacodynamic activity is expected. The modulation of activity of CYP3A and P-gp by ritonavir will be also monitored using micro dose midazolam and fexofenadine as probe substrates.

The purpose of this study is to use the Simcyp® Simulator mechanistic PBPK modeling to broaden the application field of ticagrelor, especially in HIV patients. Since PK models are often created after clinical observations, the prospective aspect of this study is of particular value as the model will be first created and then applied to an unknown clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Aged between 18 and 60 years
* BMI between 18 and 27
* Understanding of French language and able to give an inform consent.

Exclusion Criteria:

* Hypersensitivity to ticagrelor or ritonavir or any constituents of the tablets
* Concomitant diseases
* Smokers (> 20 cigarettes per day)
* Intake of any drug or food (grapefruit) that is metabolized by or can affect CYP3A or P-glycoprotein activity within the last 10 days
* Pathologies or drugs associated with an increased bleeding risk such as aspirin, non-steroidal anti-inflammatory drugs, steroids and serotonin reuptake inhibitors
* Bleeding familial history or antecedent or hemorrhagic disease
* Previous or active gastro-intestinal ulcer
* Alteration of hepatic tests (ASAT>100 U/l, ALAT >100 U/l, GGT >80 U/l, BILI > 50 μmol/l)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in AUC of ticagrelor and its metabolite from baseline | 30 min 1hr 2hr 3hr 4hr 6hr 8hr 24hr
  Venous blood samples will be taken to assess the baseline pharmacokinetic parameters of ticagrelor and its metabolite, prior to ticagrelor administration (time zero) and at the following post dosage times: 0.5, 1, 2, 3, 4, 6, 8, and 24 hours

SECONDARY OUTCOMES:
Measure of the pharmacodynamic response to ticagrelor by two platelet reactivity tests VASP and VerifyNow® P2Y12 | 4hr
  4 hours after administration of ticagrelor the pharmacodynamic, response of ticagrelor will be assessed by the VAsodilator-Stimulated Phosphoprotein Assay (VASP) and VerifyNow® P2Y12 tests
Change in P-gp phenotyping from baseline (0 min) | 30 min 1hr 2hr 3hr 4hr 6hr 8hr 24hr
  Venous blood samples will be taken to assess the P-gp phenotyping, prior to fexofenadine administration (time zero) and at the following post dosage times: 0.5, 1, 2, 3, 4, 6, 8, and 24 hours
Change in CYP3A4 phenotyping from baseline (0 min) | 1hr
  Venous blood samples will be taken to assess the CYP3A4 phenotyping, prior to midazolam administration (time zero) and at the following post dosage time: 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche Clinique, HUG, Rue Gabrielle Perret-Gentil 4, Geneva, Switzerland